CLINICAL TRIAL: NCT05895344
Title: Long-term Cognitive and Functional Impact of Proton-therapy or Modern Fractionated Radiotherapy in Cavernous Sinus Meningioma
Brief Title: Long-term Cognitive and Functional Impact of Proton-therapy or Modern Fractionated Radiotherapy in Cavernous Sinus Meningioma: An Open-label Randomized 1:1 Phase III Study
Acronym: COG-PROTON-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A00401-44
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cavernous Sinus Meningioma; Proton-therapy; Photon Radiotherapy; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Protons

STUDY DESIGN:
Intervention Model Description: Multicenter prospective comparative phase 3 randomized 1:1 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- proton-therapy (Experimental): Proton pencil-beam-scanning irradiation (50,4 Gy (RBE) in 28 fractions)
  Interventions: Radiation: Proton-therapy
- photon radiotherapy (Active Comparator): Intensity modulated radiotherapy with or without stereotactic positioning (50,4 Gy in 28 fractions)
  Interventions: Radiation: Photon radiotherapy

INTERVENTIONS:
Radiation: Proton-therapy — Proton pencil-beam-scanning irradiation (50,4 Gy (RBE) in 28 fractions)
  Arms: proton-therapy
Radiation: Photon radiotherapy — Intensity modulated radiotherapy with or without stereotactic positioning (50,4 Gy in 28 fractions)
  Arms: photon radiotherapy

SUMMARY:
Cavernous sinus meningiomas are close to optic nerve, pituitary gland, cranial nerve, and hippocampi.

The doses delivered to these structures are crucial and radiotherapy of cavernous sinus meningiomas exposes patients to late secondary effects (pituitary deficit, nerve palsy, cognitive impairment…). In 2012, Gondi reported that a dose given to 40% of the bilateral hippocampi greater than 7.3 Gy is associated with long-term impairment in list-learning delayed recall after FSRT for benign or low-grade adult brain tumors.

There is no published or recruiting prospective study evaluating the impact of proton-therapy or conventional irradiation on neurocognitive function for meningioma patients. Notably, long-term cognitive or ocular impact of these modern irradiation schemes remains poorly known. Yet, these patients had a long life-expectancy, and are at risk of developing long-term sequelae. Thus, according to its ballistic advantage, an improvement of patient functional outcomes and a reduction of neurocognitive long-term toxicity are expected if tissue sparing proton-therapy is used.

In this context, a randomized prospective study, evaluating long-term toxicity of these two irradiation modalities (Proton Therapy (PRT) and photon radiotherapy (XRT)) seems crucial to further assess proton-therapy indication for these patients.

Although literature reports excellent outcomes for intracranial meningioma patients treated by proton-therapy, none of the eight retrospective studies found in the literature used an accurate and full evaluation of long-term toxicity

ELIGIBILITY:
Inclusion Criteria:

* Cavernous sinus meningioma for which clinical target volume is larger than 3 centimeters
* Anterior skull base meningioma, invading by contiguity the cavernous sinus can be included
* Histologic proven Grade I meningioma
* Meningioma for which biopsy is not safely achievable and for which growing and imaging criteria are in favour of grade I meningioma can be included
* Age >18 years and ≤70 years
* Indication of irradiation validated by a pluridisciplinary meeting
* Adjuvant or exclusive irradiation is allowed.
* Use of conventional fractionation: 1.8Gy (RBE)/fraction
* Signed informed consent form
* WHO Performance status equal to 0 or 1
* Patient affiliated to the French social health insurance
* MoCA score ≥ cut-off of GRECOGVASC normative data (Roussel, 2016, cf annexe 1)
* Patient whose neuropsychological abilities allow to follow the requirements of the protocol

Exclusion Criteria:

* Patient with mutation in a known predisposition gene (NF-2, SMARCE-1…)
* Cerebrovascular pathology, presence of other tumors of the nervous system, congenital malformations of the nervous system, multiple sclerosis, Parkinson's disease and other dementias, organic psychosis (other than dementia), schizophrenia, and neurodegenerative disease
* Radiosurgery, hypofractionated regimen
* Other localization than cavernous sinus
* Histologic proven Grade II or III meningioma
* Patient with unadjusted antiepileptic drug
* Contraindication to MRI
* Patient with a history of brain irradiation
* Patient with a history of cancer in the last five years (excluding skin baso-cellular carcinoma)
* Pregnant/breastfeeding woman
* Any geographical conditions, social and associated psychopathology that may compromise the patient's ability to participate in the study
* Participation in a therapeutic trial for less than 30 days
* Patient deprived of freedom or under guardianship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
functional deterioration evaluated by individual neurocognitive test scores | 5 years
  Neurocognitive deterioration defined as the occurrence of cognitive impairment (a total of 5 impaired z-scores (17 z-scores for 6 different tests)

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Centre Francois Baclesse, Caen
  - Hopital d'Instruction des Armées PERCY, Clamart
  - CHU Grenoble-Alpes, Grenoble
  - Centre Guillaume le Conquerant, Le Havre
  - Centre Léon Bérard, Lyon
  - Hospices civils de Lyon, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hôpital Pitié Salpétrière, Paris
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - IUCT, Toulouse
  - Gustave Rousy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lesueur P, Clarisse B, Lequesne J, Licaj I, Feuvret L, Stefan D, Ricard D, Noel G, Balosso J, Lange M, Capel A, Durand-Zaleski I, Castera M, Legrand B, Goliot N, Hedou C, Grellard JM, Valable S. Proton therapy versus conventional radiotherapy for the treatment of cavernous sinus benign meningioma, a randomized controlled phase III study protocol (COG-PROTON-01). BMC Cancer. 2024 Dec 30;24(1):1594. doi: 10.1186/s12885-024-13353-9. PMID 39736544